CLINICAL TRIAL: NCT06684548
Title: Effect of Hip/Shoulder-Width Ratio on Sensory Blockade After Intrathecal Anesthesia for Adult Subumblical Herniorraphy
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Amr Abdelazeem Fouad, Resident doctors at Anesthesia, Intensive Care and Pain Management, Assiut University
Other Study IDs: HS W Ratio Herniorraphy
Record Dates: First submitted 2024-11-09; First posted 2024-11-12 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-11

CONDITIONS: Herniorrhaphy
Keywords: hip/shoulder-width ratio; sub umblical herniorrhaphy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

INTERVENTIONS:
Procedure: Hip/shoulder width ratio — the effect of hip/shoulder-width ratio on sensory blockade level in patients undergoing intrathecal anesthesia for subumbilical herniorrhaphy

SUMMARY:
Spinal anesthesia is a straightforward and reliable technique frequently employed in lower body surgeries, achieving adequate surgical conditions through the injection of a small amount of local anesthetic (LA) into the intrathecal space . One advantage of spinal anesthesia over general anesthesia is reduced exposure to potentially depressant drugs . However, inadequate spinal spread can result in pain and discomfort for patients and complicate surgical procedures . Consequently, anesthesiologists encounter the challenge of attaining the proper spread of spinal anesthesia for subumbilical herniorrhaphy due to individual anthropometric variations .

Approximately 25 factors have been identified that affect the spread of spinal anesthesia in the subarachnoid space for a given dose of LA . Variables that are both practically obtainable and predictive of spinal anesthesia spread can aid anesthesiologists in anticipating the extent of the block. Among the most studied factors are patient characteristics, injection techniques, patient posture, and the baricity of the LA .

Research has examined various patient variables affecting spinal anesthesia spread, including age , weight , height , gender, patient position, BMI , vertebral column length (VCL), and abdominal circumference . Body morphometrics such as the hip-shoulder width ratio (HSWR) have garnered attention for their potential impact on the distribution of anesthetic agents within the intrathecal space . Despite the well-established influence of factors like age, weight, and spinal anatomy, the specific role of HSWR in the outcomes of intrathecal anesthesia remains underexplored this study aim to To evaluate the effect of hip/shoulder-width ratio (HSWR) on sensory blockade level after intrathecal anesthesia for adult patients undergoing subumblical herniorraphy

DETAILED DESCRIPTION:
Spinal anesthesia is a straightforward and reliable technique frequently employed in lower body surgeries, achieving adequate surgical conditions through the injection of a small amount of local anesthetic (LA) into the intrathecal space . One advantage of spinal anesthesia over general anesthesia is reduced exposure to potentially depressant drugs . However, inadequate spinal spread can result in pain and discomfort for patients and complicate surgical procedures . Consequently, anesthesiologists encounter the challenge of attaining the proper spread of spinal anesthesia for subumbilical herniorrhaphy due to individual anthropometric variations .

Approximately 25 factors have been identified that affect the spread of spinal anesthesia in the subarachnoid space for a given dose of LA . Variables that are both practically obtainable and predictive of spinal anesthesia spread can aid anesthesiologists in anticipating the extent of the block. Among the most studied factors are patient characteristics, injection techniques, patient posture, and the baricity of the LA .

Research has examined various patient variables affecting spinal anesthesia spread, including age , weight , height , gender, patient position, BMI , vertebral column length (VCL), and abdominal circumference . Body morphometrics such as the hip-shoulder width ratio (HSWR) have garnered attention for their potential impact on the distribution of anesthetic agents within the intrathecal space . Despite the well-established influence of factors like age, weight, and spinal anatomy, the specific role of HSWR in the outcomes of intrathecal anesthesia remains underexplored

ELIGIBILITY:
Inclusion Criteria:

* Age 20 - 50 years old
* Both sexes
* Patients who are in risk-scoring groups I-II of the American Society of Anesthesiologists (ASA)
* Elective subumblical herniorraphy under intrathecal anesthesia

Exclusion Criteria:

* • Patient refusal

  * Patients have a contraindication for regional anesthesia, e.g. coagulopathy.
  * Failed or unsatisfactory intrathecal block.
  * Patients have a central nervous system disease (mental retardation, non-cooperated speech disorder, or psychiatric disease).
  * Patients who are under 150 cm or over 185 cm in height, or BMI >40.
  * Patients have experienced an operation lasting more than 2 h.
  * Patients with known hypersensitivity to amide local anesthetics.
  * Local injection site infection or spinal deformity.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients subjected to subumblical herniorraphy
Sampling Method: Probability Sample
Enrollment: 72 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2026-12-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
the sensory blockade level in patients undergoing intrathecal anesthesia for subumbilical herniorrhaphy. | baseline

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Ngaka TC, Coetzee JF, Dyer RA. The Influence of Body Mass Index on Sensorimotor Block and Vasopressor Requirement During Spinal Anesthesia for Elective Cesarean Delivery. Anesth Analg. 2016 Dec;123(6):1527-1534. doi: 10.1213/ANE.0000000000001568. PMID 27870737
- [Background] Fu F, Xiao F, Chen W, Yang M, Zhou Y, Ngan Kee WD, Chen X. A randomised double-blind dose-response study of weight-adjusted infusions of norepinephrine for preventing hypotension during combined spinal-epidural anaesthesia for Caesarean delivery. Br J Anaesth. 2020 Mar;124(3):e108-e114. doi: 10.1016/j.bja.2019.12.019. Epub 2020 Jan 17. PMID 31959386
- [Background] Chen M, Chen C, Ke Q. The effect of age on the median effective dose (ED50) of intrathecally administered plain bupivacaine for motor block. Anesth Analg. 2014 Apr;118(4):863-8. doi: 10.1213/ANE.0000000000000147. PMID 24651241
- [Background] Zhou QH, Xiao WP, Shen YY. Abdominal girth, vertebral column length, and spread of spinal anesthesia in 30 minutes after plain bupivacaine 5 mg/mL. Anesth Analg. 2014 Jul;119(1):203-206. doi: 10.1213/ANE.0000000000000199. PMID 24806139
- [Background] Adesope OA, Einhorn LM, Olufolabi AJ, Cooter M, Habib AS. The impact of gestational age and fetal weight on the risk of failure of spinal anesthesia for cesarean delivery. Int J Obstet Anesth. 2016 May;26:8-14. doi: 10.1016/j.ijoa.2016.01.007. Epub 2016 Feb 2. PMID 27020240
- [Background] Agegnehu AF, Gebregzi AH, Endalew NS. Review of evidences for management of rapid sequence spinal anesthesia for category one cesarean section, in resource limiting setting. Int J Surg Open. 2020;26:101-105. doi: 10.1016/j.ijso.2020.08.013. Epub 2020 Sep 3. PMID 34568612
- [Background] Shivashankar A, Rajappa GC, Sudarshan S, Madhu MM, Rao R. Evaluation of Effect of Hip/Shoulder-Width Ratio on the Sensory Level of Spinal Anesthesia - A Prospective Observational Study. Anesth Essays Res. 2022 Jan-Mar;16(1):80-83. doi: 10.4103/aer.aer_146_21. Epub 2022 Jun 27. PMID 36249129